CLINICAL TRIAL: NCT02456714
Title: Second Line Chemotherapy FOLFIRINOX in Irresectable Cholangiocarcinoma
Acronym: 4CC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Heinz-Josef Klumpen, Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: volgt
Record Dates: First submitted 2015-03-10; First posted 2015-05-28 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; FOLFIRINOX; Phase II study
MeSH Terms: conditions — Cholangiocarcinoma | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Progressive cholangiocarcinoma, second line treatment (Experimental): FOLFIRINOX
  Interventions: Drug: FOLFIRINOX

INTERVENTIONS:
Drug: FOLFIRINOX
  Other Names: Second line treatment

SUMMARY:
Cholangiocarcinoma, is a malignant gastrointestinal tumor of low incidence with a poor prognosis. Chemotherapy is the most common treatment for advanced disease. On the basis of a phase III clinical study, cisplatin plus gemcitabine is considered standard first-line treatment in advanced cholangiocarcinoma patients, but there is no established second line therapy.

Since fluorouracil and leucovorin combined with irinotecan and oxaliplatin (FOLFIRINOX) appears to be safe and demonstrated efficacy in clinical studies of advanced pancreatic cancer, colorectal cancer and a phase I study in cholangiocarcinoma, this combination could be an effective second-line treatment for patients with advanced cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of cholangiocarcinoma.
* Metastatic disease or irresectable locally advanced cholangiocarcinoma.
* Measurable disease according RECIST criteria version 1.1.
* Age from 18 to 75 year.
* WHO/ECOG performance status 0-2.
* Patients who received at least 3 cycles of gemcitabine/cisplatin in the first line.
* Adequate hematological function (WBC > 3.0 x 109/L, platelets > 100 x109/L)
* Adequate hepatic function (bilirubin ≤ 1.5 x upper normal limit (ULN); ALAT or ASAT <5x ULN in case of liver metastases and < 2.5 x ULN in absence of liver metastases.
* Adequate renal function (creatinine clearance > 60 ml/min; creatinine <120 µmol/L)
* Absence of cardiac insufficiency, chest pain (not medically controlled) and myocardial infarction in the 12 months preceding study entry.
* Signed informed consent.

Exclusion Criteria:

* Concurrent secondary malignancies or other malignancies within 3 years prior to enter this study with the exception of non-metastatic basal cell or squamous cell skin cancer or carcinoma in situ of the cervix treated by cone-biopsy or resection
* Presence of cerebral or meningeal metastases
* Contraindication to any of the substances of the planned treatment.
* History of chronic diarrhea or colorectal inflammatory conditions, or of unresolved occlusion or sub-occlusion for which symptomatic treatment is being administered
* Active infection or other serious underlying conditions which may prevent the patient from receiving the planned treatment. For example: prolonged unresolved bacterial cholangitis with destruction of bile duct branches (e.g. after endoprosthesis insertion) or two or more cholangitis in the last 6 months. Patients with other active or uncontrolled severe infection, cirrhosis or chronic active hepatitis will be excluded.
* Presence of cardiac insufficiency, unstable angina pectoris, symptomatic congestive heart, failure myocardial infarction 6 months prior to randomization, serious uncontrolled cardiac arrhythmia.
* Inclusion in another investigational clinical trial
* Women who are pregnant, breast-feeding or not using adequate contraceptive
* Age younger than 18 or older than 76 years
* Individuals under correctional supervision or guardianship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
pilot study: toxicity | 24 weeks
  number of adverse events in accordance with CTCAEv4.0
phase II: the response rate | 24 weeks

SECONDARY OUTCOMES:
pilot study: the response rate | 24 weeks
pilot study: time to progression. | 24 weeks
pilot study: the overall survival | 24 weeks
pilot study: quality of life | 24 weeks
phase II: toxicity during the treatment period and 30 days after the treatment. | 24 weeks
  number of adverse events in accordance with CTCAEv4.0
phase II: time to progression. | 24 weeks
phase II: the overall survival. | 24 weeks
phase II: quality of life | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: H.J. Klümpen, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); J. Wilmink, MD, PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic medical center Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Belkouz A, de Vos-Geelen J, Mathot RAA, Eskens FALM, van Gulik TM, van Oijen MGH, Punt CJA, Wilmink JW, Klumpen HJ. Efficacy and safety of FOLFIRINOX as salvage treatment in advanced biliary tract cancer: an open-label, single arm, phase 2 trial. Br J Cancer. 2020 Mar;122(5):634-639. doi: 10.1038/s41416-019-0698-9. Epub 2020 Jan 10. PMID 31919404
- See also: Final publication — https://www.nature.com/articles/s41416-019-0698-9.pdf